CLINICAL TRIAL: NCT00588588
Title: Bronchoscopy Versus Clinical Pulmonary Infection Score Guided Approach in Suspected Ventilator-Associated Pneumonia (VAP): Randomized Clinical Trial
Brief Title: Bronchoscopy vs. Clinical Pulmonary Infection Score Guided Approach in Suspected Ventilator-Associated Pneumonia (VAP)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to inability to get support for the study
Sponsor: Mayo Clinic (Other)
Responsible Party: Bekele Afessa, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-002660
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator associated pneumonia; Intensive Care; Antibiotics; Mortality; Length of stay
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bronchoscopy
  Interventions: Procedure: Bronchoscopy
- 2 (Active Comparator): CPIS
  Interventions: Procedure: Clinical pulmonary infection score (CPIS)

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopy procedure
  Arms: 1
Procedure: Clinical pulmonary infection score (CPIS) — Calculate CPIS
  Arms: 2

SUMMARY:
The reported incidence of ventilator associated pneumonia (VAP) is 10 to 15 per 1,000 ventilator days. VAP leads to an excess cost exceeding $40,000 per patient and is associated with a crude mortality rate as high as 76%. The clinical criteria for the diagnosis of VAP have low specificity and may lead to unnecessary antibiotic use. The Clinical Pulmonary Infection Score (CPIS) and bronchoscopic approaches lower unnecessary antimicrobial use, antimicrobial resistance, and superinfection compared to the traditional clinical criteria.

Based on the available evidence and local microbiology data, we have developed a VAP management protocol guided by CPIS or bronchoalveolar lavage (BAL) in adults with suspected VAP. These two approaches have not been compared against each other. Although the diagnostic studies in the CPIS guided approach are inexpensive and easily available, BAL has the potential to minimize the unnecessary use of antibiotics and reduce the development of drug resistant pathogens.

In this study, we propose to test the hypothesis that BAL leads to a reduction in antibiotic use compared to CPIS in patients with suspected VAP. The study design will be a randomized, clinical trial comparing CPIS versus BAL. The primary outcome measure will be antibiotic utilization. The secondary outcome measures will be mortality, morbidity, development of resistant pathogens and superinfection and infection related financial burden.

Completion of this trial will help us identify the best approach to avoid unnecessary antibiotic utilization and minimize the development of resistant pathogens (with their associated morbidity and mortality) in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Endotracheal intubation
* Suspected VAP with:
* New or progressive pulmonary infiltrates plus two of the following (In patients with pre-existing ALI or ARDS, physicians' suspicion of VAP with two of the listed criteria will be used.): Temperature > 38 C or < 36 C, WBC > 12,000/mL or < 4,000/mL, purulent endotracheal secretions.
* Patient or legally authorized representative is able to sign Informed Consent

Exclusion Criteria:

* Prison inmates
* Immunocompromised patients
* Participation in another trial conflicting with the design of the current trial
* Previous history of VAP during the same hospitalization
* Previous participation in the current study
* Concomitant non-pulmonary infection diagnosed within 3 days preceding the suspected VAP
* Patient's primary care provider does not want subject to be enrolled in the study
* Contraindications for bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
14-day antibiotic free days | Day 14 of enrolment

SECONDARY OUTCOMES:
Mortality | 28 days
Daily organ failure score | 14 days
Length of hospital stay | Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Bekele Afessa, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- [Background] Afessa B, Hubmayr RD, Vetter EA, Keegan MT, Swanson KL, Baddour LM, Cockerill FR 3rd, Peters SG. Bronchoscopy in ventilator-associated pneumonia: agreement of calibrated loop and serial dilution. Am J Respir Crit Care Med. 2006 Jun 1;173(11):1229-32. doi: 10.1164/rccm.200512-1899OC. Epub 2006 Mar 9. PMID 16528014